CLINICAL TRIAL: NCT01054417
Title: A Prospective Evaluation to Determine Laparoscopic Criteria for the Diagnosis Appendicitis During a Diagnostic Laparoscopy
Brief Title: APPEndicitis and Laparoscopic Criteria; APPEL Study
Acronym: APPEL
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, JW Haveman, Surgeon, University Medical Center Groningen
Other Study IDs: APPEL01
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Appendicitis
Keywords: Appendicitis; Laparoscopy; Appendectomy
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Slices of the appendix fixed for pathologic examnination will be retained (standard procedure).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Appendicitis: Patients with suspected appendicitis who are to be operated upon by diagnostic laparoscopy

SUMMARY:
A diagnostic laparoscopy is frequently used to confirm the diagnosis of appendicitis. However, laparoscopic criteria for determining appendicitis are not defined. If there is any doubt about the presence of an abnormal appendix, it is usually removed. However, an appendectomy of a negative appendix has a certain morbidity and for that reason it should be avoided. The purpose of this study is to establish laparoscopic criteria for the diagnosis appendicitis during diagnostic laparoscopy.

DETAILED DESCRIPTION:
The UMCG hospital protocol of suspicion of appendicitis includes a diagnostic laparoscopy. The laparoscopic inspection of the appendix is carried out according to a specific protocol. In case of appendicitis the appendix is removed laparoscopically, a normal appendix is not removed. The primary outcome of the study is: appendicitis according to pathologic examination following appendectomy, or appendicitis according to clinical follow-up in case the appendix is not removed.

The clinical diagnosis of appendicitis in the follow-up should be confirmed radiologic examination (ultrasound, CT-scan, MRI) or by a re-operation.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Patients who will undergo a diagnostic laparoscopy for suspicion of appendicitis
* No age or gender limits

Exclusion Criteria:

* Elective scheduled appendectomy
* Unable to give informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who will undergo a diagnostic laparoscopy for the clinical diagnosis appendicitis.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2009-12; Primary Completion 2011-04 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Accuracy of appendix characterization by histology or clinically | 3 months

SECONDARY OUTCOMES:
Readmission | 3 months
Re-operation | 3 months
Intra-abdominal abcess | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: JW Haveman, MD, PhD, Principal Investigator — University Medical Center Groningen, the Netherlands
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands